CLINICAL TRIAL: NCT00611299
Title: Dose-Response Study of Probiotic Bacteria Bifidobacterium Animalis Subsp. Lactis BB-12 and Lactobacillus Paracasei Subsp. Paracasei CRL-341 in Healthy Young Adults
Brief Title: Dose-Response Study of Probiotic Bacteria BB-12 and CRL-431 in Healthy Young Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BC Vcap 01
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2002-12

CONDITIONS: Cardiovascular Disease; Constipation
Keywords: Probiotics; Immune response; Blood lipids; Intestinal microflora; Tolerance
MeSH Terms: conditions — Cardiovascular Diseases; Constipation

INTERVENTIONS:
Dietary Supplement: BB-12 and CRL 431

SUMMARY:
The purpose of the study was to investigate the dose-response effect of increasing doses of Bifidobacterium animalis ssp lactis (BB-12) and Lactobacillus paracasei ssp paracasei (CRL-431) on the immune response, blood lipids, gut microflora, recovery from feces and overall tolerance in healthy young adults.

DETAILED DESCRIPTION:
The study included seventy-one healthy young vounteers, and was designed as a double-blind placebo controlled dose-response trial based on a 2 wk run-in period, a 3 wk intervention and 2 wk wash-out period. The subjects were randomly assigned into 5 groups of 15 subjects each, who were supplemented with 0, 10E8, 10E9, 10E10 or 10E10 CFU/d, respectively, og a mixture of BB-12 and CRL-431. Blood samples were collected 4 times and fecal samples 3 times. Diary reporting bowel habits and weel being was kept for all 7 weeks.

There are very few articles concerning the issue dose-response effect of probiotics.The aim of the study was to investigate the dose-response effect of increasing concentrations of probiotics on the immune response, blood lipids, composition of the gut microflora, recovery from feces and the overall tolerance.

The hypothesis was that the increasing dose would influence the immunresponse (eg incresae phagocytosis), improve blood lipid profile (eg.lower HDL-cholesterol), would be recovered in increasing concentrations in feces, would change the intestinal microfloraprofile and would be well tolerated even in high doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young individuals

Exclusion Criteria:

* GI-disease
* Colosomi
* Pregnant or lactating women
* Allergy
* Individuals receiving the following medicine: antacid, antibiotics, steroids, medicine with influence the intestinal function.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71
Dates: Start 2003-04; Study Completion 2003-11

PRIMARY OUTCOMES:
Modulation of the immune system
Influence on blood lipids
Bioavailibility of BB-12 and CRL-341
Overall tolerance
Effect on the composition of the gut microflora

CONTACTS AND LOCATIONS:
Overall Officials: Kim F Michaelsen, Prof dr med, Principal Investigator — Michaelsen KF
Locations (1):
- Department of Human Nutrition, Frederiksberg C, Denmark

REFERENCES:
- See also: probiotic dose-response influence on immunesystem, blood lipids and tolerance — http://www.probiotics.com